CLINICAL TRIAL: NCT00076245
Title: Cognitive Behavioral Approaches to Seasonal Depression
Brief Title: Cognitive Behavioral Therapy for the Treatment of Seasonal Affective Disorder (SAD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kelly Rohan, Principal Investigator, Henry M. Jackson Foundation for the Advancement of Military Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R03MH065946 (NIH); R03MH065946 (NIH); DSIR AT-AS
Record Dates: First submitted 2004-01-16; First posted 2004-01-19 (Estimated); Results first posted 2014-06-25 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Seasonal Affective Disorder; Depression
Keywords: Phototherapy
MeSH Terms: conditions — Seasonal Affective Disorder; Depression | interventions — Phototherapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 Light therapy (Experimental)
  Interventions: Behavioral: Light Therapy
- 2 Cognitive behavioral therapy (Experimental)
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)
- 3 Light therapy plus cognitive behavioral therapy (Experimental)
  Interventions: Behavioral: Light Therapy; Behavioral: Cognitive behavioral therapy (CBT)
- 4 Control (No Intervention)

INTERVENTIONS:
Behavioral: Light Therapy — Light therapy will involve exposure to bright light twice a day.
  Arms: 1 Light therapy; 3 Light therapy plus cognitive behavioral therapy
Behavioral: Cognitive behavioral therapy (CBT) — CBT attempts to change maladaptive thoughts and beliefs, and will be conducted twice a week.
  Arms: 2 Cognitive behavioral therapy; 3 Light therapy plus cognitive behavioral therapy

SUMMARY:
This study will assess the effectiveness of cognitive behavioral therapy (CBT) in treating seasonal affective disorder (SAD), commonly called the "winter blues."

DETAILED DESCRIPTION:
SAD is a condition in which people experience depression as a result of seasonal variations in sunlight. Although light therapy is a common treatment for SAD, a large proportion of people with SAD are resistant to this treatment. CBT is effective for nonseasonal depressive disorders, but its use for SAD has not been thoroughly explored. This study will determine whether CBT, alone and combined with light therapy, is as effective as light therapy alone in reducing SAD symptoms.

Participants in this study will be randomly assigned to light therapy, CBT, a combination of light therapy and CBT, or a control group (no therapy) for 6 weeks. CBT will be conducted twice a week; light therapy will be conducted twice a day. Assessments will be made before, during, and after the study treatment. Depression scales, questionnaires, and behavioral tasks will be used to assess the depressive symptoms of participants. A 6-month and 1-year follow-up visit will also be conducted. During the follow-up visits, participants will be interviewed and will complete a questionnaire and a survey.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of seasonal affective disorder (SAD)
* Willing and able to participate in the study procedures

Exclusion Criteria:

* Major psychological diagnoses other than SAD
* Current psychological or psychiatric treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2002-11; Primary Completion 2004-02 (Actual); Study Completion 2005-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly J. Rohan, PhD, Principal Investigator — Uniformed Services University of the Health Sciences (USUHS)
Locations (1):
- Uniformed Services University of the Health Sciences (USUHS), Bethesda, Maryland, United States

REFERENCES:
- See also: Association for Behavioral and Cognitive Therapies [ABCT] — http://www.abct.org/Home/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1 Light Therapy | 2 Cognitive Behavioral Therapy | 3 Light Therapy Plus Cognitive Behavioral Therapy | 4 Control
Started | 16 | 15 | 15 | 15
Completed | 16 | 15 | 15 | 14
Not Completed | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Light Therapy | 2 Cognitive Behavioral Therapy | 3 Light Therapy Plus Cognitive Behavioral Therapy | 4 Control | Total
Number analyzed (Participants) | 16 | 15 | 15 | 15 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (9.7) | 45.9 (15.5) | 43.0 (12.8) | 43.3 (7.7) | 45.0 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 15 | 14 | 12 | 55
  Male | 2 | 0 | 1 | 3 | 6
Race/Ethnicity, Customized [Number; unit: participants]
  White | 13 | 11 | 12 | 12 | 48
  Asian | 0 | 1 | 2 | 0 | 3
  African American | 2 | 2 | 1 | 2 | 7
  Hispanic | 1 | 0 | 0 | 1 | 2
  Other | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 15 | 15 | 61

OUTCOME MEASURES:

1. Primary Outcome: Scores on the Structured Interview Guide for the Hamilton Depression Rating Scale-Seasonal Affective Disorder Version
Description: The Structured Interview Guide for the Hamilton Depression Rating Scale-Seasonal Affective Disorder Version (SIGH-SAD) measures depressive symptoms on a continuous scale. Higher scores indicate worse outcome. Range of scores is 0 to 73. Generally, a score of 20 or higher is the cutoff for clinical depression.
Time Frame: Post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1 Light Therapy | 2 Cognitive Behavioral Therapy | 3 Light Therapy Plus Cognitive Behavioral Therapy | 4 Control
Number analyzed (Participants) | 16 | 15 | 15 | 15
units on a scale | 13.6 (8.8) | 13.3 (11.1) | 8.3 (5.8) | 22.6 (8.4)

2. Primary Outcome: Remission Status on Structured Interview Guide for the Hamilton Depression Rating Scale-Seasonal Affective Disorder Version (SIGH-SAD)
Description: Dichotomous Remission Status (remitted or not) at post-treatment
Time Frame: Post-treatment
Measure: Number; unit: participants
Arm/Group | 1 Light Therapy | 2 Cognitive Behavioral Therapy | 3 Light Therapy Plus Cognitive Behavioral Therapy | 4 Control
Number analyzed (Participants) | 16 | 15 | 15 | 15
participants | 8 | 6 | 11 | 3

ADVERSE EVENTS:
Arm/Group | 1 Light Therapy | 2 Cognitive Behavioral Therapy | 3 Light Therapy Plus Cognitive Behavioral Therapy | 4 Control
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No